CLINICAL TRIAL: NCT00821860
Title: Prospective Randomised Controlled Trial of Video-Assisted Thoracoscopic (VAT) Cytoreductive Pleurectomy Compared to Talc Pleurodesis in Patients With Suspected or Proven Malignant Mesothelioma
Brief Title: Video-Assisted Surgery or Talc Pleurodesis in Treating Patients With Malignant Mesothelioma
Acronym: MesoVATS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00804; PAPWORTH-MESOVATS; PAPWORTH-P00804; EU-20901; ISRCTN34321019
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Mesothelioma; Metastatic Cancer
Keywords: epithelial mesothelioma; recurrent malignant mesothelioma; sarcomatous mesothelioma; malignant pleural effusion; stage IA malignant mesothelioma; stage IB malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma; stage IV malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Neoplasm Metastasis; Solitary Fibrous Tumor, Pleural; Pleural Effusion, Malignant | interventions — Talc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo video-assisted thoracoscopic cytoreductive pleurectomy either at the time of biopsy or after confirmation of biopsy results.
  Interventions: Procedure: therapeutic videothoracoscopy
- Arm II (Active Comparator): Patients undergo talc pleurodesis via an indwelling intercostal chest drain or via thoracoscopy either at the time of biopsy or after confirmation of biopsy results.
  Interventions: Other: talc; Procedure: therapeutic thoracoscopy

INTERVENTIONS:
Other: talc — Talc pleurodesis
  Arms: Arm II
Procedure: therapeutic thoracoscopy — Talc pleurodesis via thoracoscopy
  Arms: Arm II
Procedure: therapeutic videothoracoscopy — Video-assisted thoracoscopic pleurectomy
  Arms: Arm I

SUMMARY:
RATIONALE: Video-assisted surgery to remove part of the tissue layer covering the inside of the chest cavity may be effective in treating pleural effusion and cause less damage to normal tissue. Talc pleurodesis may keep fluid from building up in the chest cavity. It is not yet known which therapy is more effective in treating pleural effusion caused by malignant mesothelioma.

PURPOSE: This randomized phase III trial is studying video-assisted surgery to see how well it works compared with talc pleurodesis in treating patients with malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effectiveness of video-assisted thoracoscopic cytoreductive pleurectomy vs talc pleurodesis, in terms of 1-year survival, in patients with suspected or proven malignant mesothelioma.

Secondary

* Compare the control of pleural effusion in these patients.
* Compare procedure-related complications in these patients.
* Compare the symptoms and quality of life of these patients at 3, 6, and 12 months after treatment.
* Compare the length of hospital stay for these patients.
* Compare the exercise tolerance of these patients at 3, 6, and 12 months after treatment.
* Determine the cost to the health service, in terms of resources used for procedures, hospital bed usage, and cost of primary and secondary care over 12 months.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (high vs low). Patients are randomized to 1 of 2 treatment arms.

* Arm I (video-assisted thoracoscopic [VAT] cytoreductive pleurectomy): Patients undergo VAT cytoreductive pleurectomy either at the time of biopsy or after confirmation of biopsy results.
* Arm II (talc pleurodesis): Patients undergo talc pleurodesis via an indwelling intercostal chest drain or via thoracoscopy either at the time of biopsy or after confirmation of biopsy results.

Quality of life, complications, and resource use are assessed at baseline and at 1, 3, 6, and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed or suspected mesothelioma

  * Any subtype allowed
* Pleural effusion must be present

PATIENT CHARACTERISTICS:

* Clinically fit and suitable for video-assisted thoracoscopic cytoreductive pleurectomy
* Prior malignancy allowed provided it no longer requires treatment AND patient has a confirmed diagnosis of mesothelioma

PRIOR CONCURRENT THERAPY:

* No prior attempted pleurodesis by any approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2003-09; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Survival at 1 year after treatment | 1 year

SECONDARY OUTCOMES:
Control of pleural effusion | 1 year
Complications, including need for more surgery, persistent air leak requiring pleural intubation for > 10 days, and hospital stay for > 12 days | 1 year
Symptoms and quality of life as assessed by the EuroQol questionnaire | 0, 1, 3, 6 12 months
Length of hospital stay | 1 year
Exercise tolerance | 0, 1, 3, 6 12 months
Cost to the health service, in terms of resources used for procedures, hospital bed usage, and cost of primary and secondary care over 12 months | 0, 1, 3, 6 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Winter, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Basildon University Hospital, Basildon, England
  - Papworth Hospital, Cambridge, England
  - Glenfield Hospital, Leicester, England
  - Guy's Hospital, London, England
  - Royal Hallamshire Hospital, Sheffield, England

REFERENCES:
- [Derived] Rintoul RC, Ritchie AJ, Edwards JG, Waller DA, Coonar AS, Bennett M, Lovato E, Hughes V, Fox-Rushby JA, Sharples LD; MesoVATS Collaborators. Efficacy and cost of video-assisted thoracoscopic partial pleurectomy versus talc pleurodesis in patients with malignant pleural mesothelioma (MesoVATS): an open-label, randomised, controlled trial. Lancet. 2014 Sep 20;384(9948):1118-27. doi: 10.1016/S0140-6736(14)60418-9. Epub 2014 Jun 16. PMID 24942631